CLINICAL TRIAL: NCT06743191
Title: Feasibility of Delivering a Digital Health Intervention to Improve Food Access and Dietary Quality Among Adults With Hypertension
Brief Title: Delivering a Digital Health Intervention to Improve Food Access and Dietary Quality Among Adults With Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB00447049; R21NR021041 (NIH)
Record Dates: First submitted 2024-12-16; First posted 2024-12-19 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Hypertension
Keywords: Digital Health; Health Behavior; Nutrition; Hypertension; Food Access
MeSH Terms: conditions — Hypertension; Health Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Assess the feasibility of Access Nourish in a 4-month study among adults with hypertension li (Experimental): All participants will be prospectively assigned to receive a behavioral intervention that includes skills training, nutrient goal setting, self-monitoring via dietary tracking, personalized text message feedback, and adaptive health coaching. Participants will also receive a membership to Instacart+ and weekly grocery list recommendations from a health coach. All intervention will be delivered remotely using smartphone technology.
  Interventions: Behavioral: Access Nourish

INTERVENTIONS:
Behavioral: Access Nourish — A total of 65 participants with hypertension and low access to high quality food will be enrolled to test the feasibility of using commercially available grocery delivery services, simultaneous to a robust behavioral intervention, to improve adherence to the DASH eating pattern. The behavioral intervention will include skills training, nutrient goal setting, self-monitoring via dietary tracking, personalized text message feedback, and adaptive health coaching. Participants will also receive a membership to Instacart+ and weekly grocery list recommendations from a health coach. Participants will be able to complete all intervention components via smartphone. The intervention period for participants will be 4 months.

SUMMARY:
A total of 65 participants with hypertension and low access to high quality food will be enrolled to test the feasibility of using commercially available grocery delivery services, simultaneous to a robust behavioral intervention, to improve adherence to the Dietary Approaches to Stop Hypertension (DASH) eating pattern. The behavioral intervention will include skills training, nutrient goal setting, self-monitoring via dietary tracking, personalized text message feedback, and adaptive health coaching. Participants will also receive a membership to Instacart+ and weekly grocery list recommendations from a health coach. The primary outcome will be indicators of feasibility, including acceptability, demand, implementation and practicality and adaption. Change in DASH adherence and blood pressure will also be evaluated. The intervention period for participants will be 4 months.

ELIGIBILITY:
Inclusion Criteria:

* Adult 18 years of age or older
* Has hypertension, defined as a systolic BP of 130-159 mmHg and/or diastolic BP of 80-99 mmHg, whether or not taking hypertension medication.
* Resides in a census tract defined as low access by the United States Department of Agriculture (USDA)
* Resides in a zip code serviced by the grocery delivery app
* BMI 18.5 kg/m2+
* Has a smartphone with a data plan
* Willing to receive daily text messages
* Can participate in online videoconference visits
* Can read and write in English

Exclusion Criteria:

* Participating in another related research study
* Cardiovascular disease event in the last 6 months
* Active cancer
* Recent hospitalization due to psychiatric condition or event
* Pregnancy or planned during the study period
* BMI 37 kg/m2 or higher
* Documented dementia
* On kidney dialysis
* Instructed to eat a low potassium diet
* Planned or recent bariatric surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2025-02-27 (Actual); Primary Completion 2025-12-18 (Actual); Study Completion 2025-12-18 (Actual)

PRIMARY OUTCOMES:
Feasibility as assessed by survey | 4 months
  Feasibility will be measured by a 23-item questionnaire used to assess participants' perceptions of the feasibility, usability, acceptability, practicality, and satisfaction with the intervention. Each item is rated on a 5-point Likert scale, with higher scores indicating greater feasibility and acceptability. The survey evaluates key components of the program, including grocery lists, grocery delivery, health coaching, and app-based tracking.

SECONDARY OUTCOMES:
Change in DASH Score as assessed by the Automated Self-Administered 24-hour (ASA24) | Baseline and 4 months
  Participants will enter dietary intake online via the National Cancer Institute's Automated Self-Administered 24-hour (ASA24) Dietary Assessment tool. DASH dietary nutrients are then converted into a score. Scores ranged from 0 to 9 where a higher score indicates better adherence to the DASH dietary pattern. Change in DASH score = 4-month DASH score - Baseline DASH score.
Change in Systolic Blood Pressure | Baseline and 4 months
  Systolic blood pressure will be measured in millimeters of mercury (mmHg) using the upper arm three times at 1-minute intervals after 5 minutes of quiet sitting. The final 2 measurements will be averaged together for analysis. Change in systolic blood pressure = 4-month systolic blood pressure - Baseline systolic blood pressure.
Change in Diastolic Blood Pressure | Baseline and 4 months
  Diastolic blood pressure will be measured in millimeters of mercury (mmHg) using the upper arm three times at 1-minute intervals after 5 minutes of quiet sitting. The final 2 measurements will be averaged together for analysis. Change in diastolic blood pressure = 4-month diastolic blood pressure - Baseline diastolic blood pressure.

CONTACTS AND LOCATIONS:
Overall Officials: Hailey Miller, RN, PhD, Principal Investigator — Johns Hopkins University; Gary Bennett, PhD, Principal Investigator — Duke University
Locations (1):
- Johns Hopkins, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No